CLINICAL TRIAL: NCT01131065
Title: Efficacy and Safety of Niuliva® for the Prevention of Hepatitis B Virus Recurrence in Newly Orthotopic Liver Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IG0907
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B; Liver Transplantation
Keywords: Hepatitis B; HBV; Orthotopic liver transplantation; Liver transplantation; Recurrence; Reinfection; Protective titers; HBsAb; Hepatitis B virus immune globulin; Niuliva
MeSH Terms: conditions — Hepatitis B; Recurrence; Reinfection | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatitis B immune globulin (Experimental): Treatment group (newly liver transplanted subjects due to HBV induced liver disease)
  Interventions: Drug: Hepatitis B immune globulin

INTERVENTIONS:
Drug: Hepatitis B immune globulin — Daily doses of 10,000 IU of intravenous hepatitis B immune globulin during the first week post-transplantation (anhepatic phase + days 1-7), followed by weekly and monthly doses of 5,000 IU during weeks 2,3, and 4 and months 2,3,4,5,6,7,8,9,10,11 and 12, respectively.
  Other Names: Niuliva

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy, safety, and tolerability of Niuliva (Hepatitis B virus immune globulin) in the prophylaxis of hepatitis B virus (HBV) reinfection in patients submitted to liver transplantation due to HBV-induced liver disease by reaching and maintaining certain hepatitis B antibody (HBsAg) levels considered as protective during the first six and twelve months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Patients from 18 to 70 years of age (both included).
* Serum HBV DNA-negative determined by DNA PCR-amplification assay just prior to anhepatic phase visit.
* Serum HBeAg negative just prior to anhepatic phase visit.
* Patients who are to undergo liver transplantation due to liver disease associated to HBV.
* The patient agrees to participate and comply with all the aspects of the protocol, including blood sampling, for the total duration of the study.
* Signed informed consent.

Exclusion Criteria:

* Patients who have already experienced a liver transplantation even for reasons not related to HBV infection.
* Patients with unknown serum HBV replication status (data on HBeAg and HBV DNA).
* Patients with known allergies to any component of Niuliva®.
* History of serious adverse events (SAEs) or frequent adverse events (AEs) related to the administration of human blood-derived products.
* Patient with unknown viral status for HCV, HAV, HIV type 1 and type 2
* Patients with selective IgA deficiency.
* Any haemostatic abnormality contraindicating i.v. injection according to the investigator's judgment.
* Patient suffers from any acute or chronic medical, surgical or psychiatric condition or laboratory abnormality that may increase the risk associated with the study participation or investigational product administration, or may interfere with the interpretation of the study results.
* Known abuse of alcohol, drugs or other chemical substances; or has done so in the past 6 months.
* Breast-feeding women or pregnant women at the time of inclusion or who are expecting to be pregnant within the next 7 months after inclusion.
* Subject has participated in any other investigational study within the last 3 months.
* Existing possibility that the patient may be treated with other products containing specific anti-hepatitis B immunoglobins (other than Niuliva®) in a period of 13 months.
* Subject is incapable of giving consent personally.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - A.O.U. Policlinico Università di Modena e Reggio Emilia, Modena, Modena
  - Az. Ospedaliera Universitaria di Padova, Padua, Padova
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - Az. Ospedaliera S.Giovanni Battista di Torino, Torino, Torino

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen subjects (newly liver transplanted due to HBV induced liver disease) were screened in the study, all received the study medication, and all completed the clinical study.
  First subject enrolled - 26 July 2010 Last subject completed - 16 June 2014
Groups:
- Hepatitis B Immune Globulin: Treatment group
  Hepatitis B immune globulin: Daily doses of 10,000 IU of intravenous hepatitis B immune globulin during the first week post-transplantation (anhepatic phase + days 1-7), followed by weekly and monthly doses of 5,000 IU during weeks 2,3, and 4 and months 2,3,4,5,6,7,8,9,10,11 and 12, respectively.
Period: Overall Study
Arm/Group | Hepatitis B Immune Globulin
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hepatitis B Immune Globulin
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — 18 to 70 years of age (inclusive)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 15
Alcohol consumption - abstemious [Number; unit: participants] | 15
Height [Mean (Standard Deviation); unit: centimeters] | 170.33 (8.08)
Weight [Mean (Standard Deviation); unit: kilogram] | 73.73 (12.05)
Hepatitis history [Number; unit: participants]
  Has chronic HBV | 15
  Has fulminant HBV | 0

OUTCOME MEASURES:

1. Primary Outcome: HBV Recurrence
Description: HBV recurrence is measured by seroconversion or reappearance of HBsAg and HBV DNA positivity
Time Frame: First six and twelve months after liver transplantation
Measure: Number; unit: participants
Arm/Group | Hepatitis B Immune Globulin
Number analyzed (Participants) | 15
participants
  Six Months | 0
  Twelve Months | 0

2. Primary Outcome: HBsAb Pre-infusion Levels (Trough Levels Before Each Niuliva Administration)
Time Frame: Days 3 to 7, Weeks 2 to 4, Months 2 to 6, and Months 7 to 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Hepatitis B Immune Globulin
Number analyzed (Participants) | 15
IU/L
  Day 3 | 764.7 (375.91)
  Day 4 | 910.7 (282.39)
  Day 5 | 969.6 (96.13)
  Day 6 | 1000.0 (0.00)
  Day 7 | 1000.0 (0.00)
  Week 2 | 1073.6 (244.21)
  Week 3 | 945.2 (250.38)
  Week 4 | 1029.2 (175.21)
  Month 2 | 592.5 (260.14)
  Month 3 | 439.2 (218.22)
  Month 4 | 398.1 (272.68)
  Month 5 | 351.9 (179.01)
  Month 6 | 369.0 (182.75)
  Month 7 | 277.7 (89.14)
  Month 8 | 304.3 (50.24)
  Month 9 | 266.0 (34.70)
  Month 10 | 301.0 (61.99)
  Month 11 | 273.3 (117.93)
  Month 12 | 284.3 (137.47)

3. Secondary Outcome: Safety and Tolerance
Description: Safety and tolerance to the product administration will be measured by the detection of adverse events or clinically relevant changes in vital signs.
Time Frame: During and after each product administration (during the 12 month treatment period)
Measure: Number; unit: participants
Arm/Group | Hepatitis B Immune Globulin
Number analyzed (Participants) | 15
participants | 15

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 12 month following orthotopic liver transplant.
Description: The duration of treatment was 6 months after which subjects were offered the option to be treated for an additional 6 months (12 months total).
Arm/Group | Hepatitis B Immune Globulin
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis B Immune Globulin (N=15)
Pyrexia (General disorders) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 1 (1)
Liver transplant rejection (Immune system disorders) | 1 (1)
Liver function tests abnormal (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis B Immune Globulin (N=15)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Localized intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Kell blood group positive (Investigations) | 1 (1)
Pharyngeal culture positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Hypokinesis (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Sleep disorders (Psychiatric disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsor's request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsor's request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor's Inventions.